CLINICAL TRIAL: NCT00004004
Title: A Phase I/II Study of Oral Procarbazine in the Treatment of Recurrent High Grade Astrocytomas
Brief Title: Procarbazine in Treating Patients With Recurrent Brain Tumor
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New Approaches to Brain Tumor Therapy Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067214; NABTT-9901; JHOC-NABTT-9901
Record Dates: First submitted 1999-11-01; First posted 2003-08-20 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2007-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Gliosarcoma | interventions — Procarbazine

INTERVENTIONS:
Drug: procarbazine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of procarbazine in treating patients who have progressive or recurrent astrocytoma, oligodendroglioma, or glioblastoma multiforme following treatment with radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of oral procarbazine when administered to patients with recurrent glioma receiving or not receiving anticonvulsants metabolized by the P450 hepatic enzyme complex.
* Determine the pharmacokinetics of oral procarbazine, including any effects of hepatic enzyme inducing drugs, in these patients.
* Assess the response rate to procarbazine in these patients.
* Evaluate this regimen in terms of overall survival and duration of disease free survival in these patients.
* Evaluate the toxicity of this regimen in these patients.

OUTLINE: Phase I of this study is a dose escalation study. Patients are stratified according to concurrent use of anticonvulsant drugs that induce cytochrome P450 (yes vs no drugs or modest-induction drugs).

* Phase I: Patients receive oral procarbazine once daily for 5 days. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of oral procarbazine until the maximum tolerated dose (MTD) is determined.

* Phase II: Once the MTD is determined, patients receive procarbazine as in Phase I.

Patients are followed every 2 months until death.

PROJECTED ACCRUAL: A total of 24-35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven malignant glioma of one of the following types:

  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Glioblastoma multiforme
* Progressive or recurrent disease after radiotherapy with or without chemotherapy
* Measurable disease by serial MR or CT

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Greater than 2 months

Hematopoietic:

* Absolute neutrophil count at least 1500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGPT/SGOT no greater than 4 times upper limit of normal

Renal:

* Creatinine no greater than 1.7 mg/dL

Other:

* No serious concurrent infection
* No other illness that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior malignancy within the past 5 years except curatively treated basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent filgrastim (G-CSF) during the first course

Chemotherapy:

* See Disease Characteristics
* No more than 1 prior chemotherapy regimen
* At least 3 weeks since prior chemotherapy (at least 6 weeks since prior nitrosoureas)
* No more than 2 prior courses of carmustine or lomustine and no greater than 460 mg/m2 or 220 mg/m2, respectively
* No prior procarbazine

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 3 months since prior radiotherapy

Surgery:

* Prior surgery allowed

Other:

* Recovered from toxicity of prior therapy
* At least 10 days since prior anticonvulsants for patients in Arm II
* No concurrent investigational agents
* No concurrent ethanol, ephedrine, isoproterenol, epinephrine, tricyclic antidepressants, paragyliline, narcotic analgesics, antihistamines, phenothiazines, hypotensives, or barbiturates
* At least 14 days since prior antidepressants (e.g., SSRI and/or MAO inhibitor)
* Must avoid foods high in tyramine (i.e., dark beer, wine, yogurt, cheese, bananas)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-07; Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A. Grossman, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (10):
- United States (10):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Result] He X, Batchelor TT, Grossman S, Supko JG; New Approaches to Brain Tumor Therapy (NABTT) CNS Consortium. Determination of procarbazine in human plasma by liquid chromatography with electrospray ionization mass spectrometry. J Chromatogr B Analyt Technol Biomed Life Sci. 2004 Jan 25;799(2):281-91. doi: 10.1016/j.jchromb.2003.10.061. PMID 14670747